CLINICAL TRIAL: NCT03669926
Title: Digital Breast Tomosynthesis - The Future Screening Tool for Breast Cancer?
Brief Title: The Tomosynthesis Trial in Bergen - Part 2
Acronym: To-Be 2
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Norwegian Institute of Public Health (Other Government)
Collaborators: Haukeland University Hospital (Other); University of Oslo (Other); Norwegian Cancer Society (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 17/209; 190184-2017 (Other Grant/Funding Number: Norwegian Cancer Society)
Record Dates: First submitted 2018-09-03; First posted 2018-09-13 (Actual); Last update posted 2024-08-28 (Actual); Status verified 2023-09

CONDITIONS: Breast Neoplasms
Keywords: Diagnostic Imaging; Mammography; Tomosynthesis; Breast cancer screening; Subsequent screening; Cancer detection; Cost effectiveness; Early performance measures; Interval cancer
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- DBT+SM (Other): Digital Breast Tomosynthesis+synthetic mammography (DBT+SM) All women are screened with DBT+SM. All examinations are independently double read. Consensus used to decide whether or not to recall.
  Interventions: Radiation: Digital Breast Tomosynthesis+synthetic mammography

INTERVENTIONS:
Radiation: Digital Breast Tomosynthesis+synthetic mammography — Two-view tomosynthesis performed with GE Senographe Pristina.
  Other Names: DBT+SM

SUMMARY:
The aim of the study is to compare early performance measures and economic aspects of organized breast cancer screening for women screened using digital breast tomosynthesis+synthetic mammography (DBT+SM) to women with a prior DBT+SM or digital mammography (DM) from To-Be 1 (NCT02835625).

DETAILED DESCRIPTION:
Digital breast tomosynthesis (DBT) is a new "three-dimensional" screening tool for breast cancer, claimed to be superior to standard two-dimensional (2D) digital mammography (DM) based on results of lower or similar recall rate, and a 30-50% higher rate of screen-detected breast cancer for DBT compared to DM.

The Bergen Tomosynthesis Trial (To-Be) is a randomized controlled trial investigating whether DBT, including synthetic mammography (SM), is superior for breast cancer screening to DM (ClinicalTrials.gov Identifier: NCT02835625) - hereafter referred to as To-Be 1. The study is run as part of BreastScreen Norway (inviting women aged 50-69 to screening every two years). It started in October 2015 and finished recruitment in December 2017, after two years - one screening round - of data collection.

Results from To-Be 1 will fill some of the knowledge gaps regarding DBT+SM in screening. However, running To-Be 1 and recent publications on the topic have identified additional challenges and new evidence gaps that are important to address before DBT can be considered for use in organized screening. Thus, the To-Be trail will be extended with five more year (To-Be 2), consisting of one additional screening round (two years) where all women in the study population are screened with DBT+SM with a three year follow-up.

To investigate the effect of subsequent screening with DBT+SM all women attending mammography screening in Bergen in 2018 and 2019 will be screened with DBT+SM. To-Be 2 is a prospective cohort study targeting 32 000 women, and all women attending screening will be asked if they are willing to take part in the study after receiving written and oral information about the study. Women willing to participate in the study will sign an informed consent form. We expect a participation rate of 90%. The participating women will be screened with DBT+SM. Women not willing to participate in the study will be screened with DM, and not included in our study.

Continuing To-Be 1 with To-Be 2 is the only opportunity to get information on women subsequently screened with DBT+SM, that have a prior DBT+SM or DM based on random allocation. This will also allow the investigators to analyze data on interval breast cancer among women screened with DBT+SM after DBT+SM and with DBT+SM after DM in To-Be 1 in 2020.

The investigators aim to address the following topics and research questions:

Part I: Early performance measures for screening with DBT+SM after DBT+SM, and DBT+SM after DM.

Part II: Interval breast cancer following screening with DBT+SM versus DM, focusing on interval breast cancers identified among women screened in To-Be 1.

Part III: Missed and true screen-detected and interval breast cancer in mammographic screening with DBT+SM versus DM.

Part IV: Expected and experienced discomfort and pain in DBT+SM by compression force and pressure.

Part V: Economic evaluation of continuous use of DBT.

ELIGIBILITY:
Inclusion Criteria:

* Written, informed consent to participation

Exclusion Criteria:

* No written, informed consent to participation
* Breast implants

Ages: 48 Years to 71 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — Only women are invited to breast cancer screening in BreastScreenn Norway.
Enrollment: 31082 (Actual)
Dates: Start 2018-01-01 (Actual); Primary Completion 2020-06-30 (Actual); Study Completion 2023-06-30 (Actual)

PRIMARY OUTCOMES:
Compare rates of screen detected breast cancer after subsequent screening with DBT+SM after DBT+SM versus screening with DBT+SM after prior DM, as performed in a population based screening program. | 48 months from start up of the trial
  Rate of screening detected breast cancer, among those screened

SECONDARY OUTCOMES:
Compare recall rates after subsequent screening with DBT+SM after DBT+SM versus screening with DBT+SM after prior DM, as performed in a population based screening program. | 48 months from start up of the trial
  Rate of recalled women due to mammographic findings, among those screened
Positive predictive value of recalls after subsequent screening with DBT+SM after DBT+SM versus screening with DBT+SM after prior DM, as performed in a population based screening program. | 48 months from start up of the trial
  Rate of breast cancer cases among those recalled
Prognostic and predictive tumor characteristics for screening detected breast cancer after subsequent screening with DBT+SM after DBT+SM versus screening with DBT+SM after prior DM, as performed in a population based screening program. | 48 months from start up of the trial
  Distribution of characteristics among the women diagnosed with breast cancer
Rate of interval breast cancer following screening with DBT+SM after DBT+SM versus screening with DBT+SM after prior DM, as performed in a population based screening program. | 48 months from start up of the trial
  Rates and prognostic and predictive tumor characteristics of interval cancer among women screened in To-Be 1, stratified by mammographic density.
Rate of missed and true screen-detected and interval breast cancer in mammographic screening with DBT+SM versus DM. | 24-48 month after start up of the trial
  Retrospective review of prior and actual mammograms from women with interval and screen-detected breast cancers detected in To-Be 1 and 2, respectively.
Economical aspects of continuous use of DBT+SM | 48 months from start up of the trial
  Estimation of the financial impact of running a screening program with DBT+SM in an everyday setting.
Comparing interpretation times to investigate possible learning effects when reading DBT+SM in two consecutive screening rounds | 48 months from start up of the trial
  Evaluation of difference in interpretation time for subsequent versus prevalent DBT+SM screens
Assessing degree of experienced and expected pain in DBT+SM screening by compression pressure using questionnaire | 6 to 48 months after start up of the trial
  Explore whether individualized, standardized compression pressure influences women's screening experiences using a numeric rating scale (0 "No discomfort/pain" to 10 "Very much discomfort/pain"). Drafting of the questionnaire is in progress.

CONTACTS AND LOCATIONS:
Overall Officials: Solveig Hofvind, Professor, Principal Investigator — Norwegian Institute of Public Health
Locations (1):
- Cancer Registry of Norway, Oslo, Norway

IPD SHARING:
Plan to Share IPD: No
We will not share the data outside the project group